CLINICAL TRIAL: NCT05137652
Title: Comparison Between One-Needle Vs Three-Needle Technique for Lumbar Radiofrequency Medial Branch Denervation in Pain Management of Low Back Pain Due to Facet Joint Arthritis
Brief Title: One-Needle Vs Three-Needle Radiofrequency in Low Back Pain Due to Facet Joint Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amani Hassan Abdel-Wahab, Professor of anesthesia, ICU and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB:17200664
Record Dates: First submitted 2021-09-18; First posted 2021-11-30 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Lumbar Facet Joint Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): single needle approach for 40 patients in which nerve is traditionally been targeted.
  Interventions: Device: Radiofrequency ablation of medial nerve using single needle approach
- Study group (Experimental): 40 patients will receive the three needle approach.
  Interventions: Device: Radiofrequency ablation of medial nerve using three needle approach

INTERVENTIONS:
Device: Radiofrequency ablation of medial nerve using single needle approach — The primary outcome is to study the efficacy of the described technique which creates a lesion that we estimate to be 11.0-mm wide and 11.6-mm long along the course of the medial branch adjacent to the SAP ensuring adequate coverage and treatment using VAS score. Responder status was defined as a 30% or greater improvement in VAS pain score from the pre-procedural VAS pain score. Outcomes were summarized by means and standard deviations for continuous outcomes, and frequencies (%) for categorical outcomes.
  Other Names: Control group
  Arms: Control group
Device: Radiofrequency ablation of medial nerve using three needle approach — The primary outcome is to study the efficacy of the described technique by maximizing the lesion size (compared to control group) along the course of the medial branch adjacent to the SAP ensuring adequate coverage and treatment using VAS score.
  Other Names: Study group
  Arms: Study group

SUMMARY:
Failure of RFA has been attributed to technical failure of coagulating the nerve or coagulation of a minimal section of the nerve, allowing for early reinnervation. Consequently, increasing the success rate and duration of relief may require techniques that increase the likelihood of successful nerve ablation over a relevant distance by maximizing lesion size.

DETAILED DESCRIPTION:
Low back pain (LBP) is more accurately called lumbago or lumbosacral pain, which is defined as discomfort, tension, or stiffness below the costal margin and above the inferior gluteal folds. In Egypt, patients with LBP constituted a high percentage of patients seeking medical care at outpatient's clinics reaching about 48% making it one of the most common causes of disability in the working population. no large-scale retrospective studies have investigated long-term clinical predictors of success in individuals receiving radiofrequency ablation (RFA) of the medial branches for facet joint arthropathy. Employees who are unable to work due to back pain spend a significant amount of time on sick leave, which impacts the productivity in the work place. Risk factors for LBP are multifactorial, including exercise, obesity, smoking, age, and sex, and these can be grouped together as individual fa pctors. Low back pain can arise from multiple anatomic locations: the intervertebral discs that are positioned between the vertebral bodies of the spine, the facet joint, but also non bony structures such as the paravertebral muscles, ligaments, and fascia. Postmortem studies have revealed that intervertebral discs and facet joints exhibit the greatest degree of degeneration within the spine, thus indicating the potential role of these structures in causing low back pain. In patients with a structural cause of low back pain, up to 40% of cases likely arise from the lumbar facet joints. The etiology of lumbar facet-joint pain is thought to be stress and trauma to the joint, which subsequently leads to inflammation of the joint capsule. Treatment options for facet arthropathy range from conservative management with medications and physical therapy to interventional management, including facet-joint injections and radiofrequency ablation (RFA) of the medial branches of the posterior rami to the facet joints. RFA of the medial branches of the dorsal rami is thought to be the most effective interventional treatment for facet joint pain and has been reported to relieve pain for 6 months to 1 year in 60% of patients. Although providing benefit in a significant proportion of patients, there remains a group of patients who do not experience any pain relief from RFA or experience only benefit from the ablation for a short period.

Failure of RFA has been attributed to technical failure of coagulating the nerve or coagulation of a minimal section of the nerve, allowing for early reinnervation. Consequently, increasing the success rate and duration of relief may require techniques that increase the likelihood of successful nerve ablation over a relevant distance by maximizing lesion size.

The aim of this technical note is to detail a two-needle approach to lumbar medial branch RF denervation to maximize lesion size along the course of the medial branch nerve.

VAS scores were based on self-reported measures of lumbar back pain and were recorded as a continuum between 2 ends of a scale, with "no pain" corresponding to the left end of the scale (0 cm) and "worst pain" corresponding to the right end of the scale (10 cm). The VAS is a validated, subjective tool to measure both acute and chronic pain. Pre-procedural VAS pain scores were documented prior to the lumbar RFA procedure (pre-VAS) and during the following time points after lumbar medial branch RFA was performed: short-term (1-week to 1-month), 3-month, 6-month, and 1-year visits.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 18-60 yrs who are complaining of chronic lower back pain due to lumbar facet joint arthritis not responded to medical treatment for more than 6 months.
* Failed back surgery syndrome without instrumentation.

Exclusion Criteria:

* Patient or relative in charge refusal.
* Associated lumbar disc prolapse.
* Negative diagnostic test.
* Contraindication for radiological exposure as pregnancy and osteoporosis.
* Inability to lie in a prone position.
* Failed back surgery syndrome with previous instrumentation insertion
* Contraindications for regional techniques

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Improvement in VAS pain score. | 24 months
  Responder status was defined as a 30% or greater improvement in pain Visual Analogue Score from the pre-procedural pain VAS score.
  The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult diseases including low back pain.
  The pain VAS originated from continuous visual analog scales developed in the field of psychology to measure well-being. the first reported use of the VAS pain scale was with the descriptor extremes "no pain at all" and "my pain is as bad as it could possibly be" in patients with a variety of conditions.

SECONDARY OUTCOMES:
Decrease the rate of recurrence of low back pain due to facet arthritis | 24 months
  regarding low back pain of lumbar facet arthritis, the secondary outcome is to decrease the rate of recurrence, the need of prolonged periods of adjuvant pharmacological treatment, the need of future surgical intervention or even the need of further sessions of radiofrequency ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abbas Youssef, Professor, Study Director — Professor of anesthesia, intensive care and Pain Relief, Assiut University; Abdelraheem Elawamy, Ass. prof., Study Director — Associate Professor of anesthesia, intensive care and Pain Relief, Assiut University
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No